CLINICAL TRIAL: NCT06783439
Title: Ultrasonographic Evaluation of the Sciatic Nerve in Patients With Piriformis Syndrome
Acronym: Sciatica
Status: Recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Busra Sezer Kıral, medical doctor, Istanbul University - Cerrahpasa
Other Study IDs: 2024-69; Istanbul PMR (Other: Istanbul PMR Training and Research Hospital)
Record Dates: First submitted 2025-01-07; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Sciatica; Piriformis Muscle Syndrome
Keywords: Piriformis Muscle Syndrome; Sciatica
MeSH Terms: conditions — Sciatica; Piriformis Muscle Syndrome | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- symptomatic hip: Patients aged between 18 and 70 years with unilateral hip and/or leg pain, positive FAIR (flexion, adduction, internal rotation) test, and tenderness to palpation in the PM will be included in our study.
  Interventions: Other: Ultrasound
- asymptomatic hip: Patients aged between 18 and 70 years with unilateral hip and/or leg pain, positive FAIR (flexion, adduction, internal rotation) test, and tenderness to palpation in the PM will be included in our study.
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Ultrasound — The ultrasound probe will be placed parallel to the body of the piriformis muscle on an imaginary line drawn from the sacrum to the greater trochanter of the femur. This area is also the sensitive area of the patients during the examination with pressure, and when the US probe is in this position, the subcutaneous fat tissue, gluteus maximus muscle, piriformis muscle, and the upper and lower borders of the sciatic nerve will be displayed in order from superficial to deep. First, the maximum thickness of the piriformis muscle body will be measured, then the thickness of the sciatic nerve will be measured, and the same measurements will be applied to the patient's asymptomatic hip, and the measurements will be recorded.

SUMMARY:
Piriformis syndrome (PS) is defined as a neuropathy of entrapment resulting from compression and irritation of the sciatic nerve at the level of the piriformis muscle (PM) at the pelvic outlet, causing sciatica radiating to the leg. The neuropathic component of PS is the compression of the sciatic nerve in or around the PM, while the primary cause of the somatic component is myofascial pain of the PM. PS accounts for 6-8% of all hip and sciatic pain cases. It is more common in middle-aged patients, and the most common etiological cause is trauma. There are various methods for the diagnosis of Piriformis Syndrome. Clinically, tenderness on palpation of the PM is the most common symptom. The FAIR test (passive flexion abduction and internal rotation of the hip), the Freiberg test (forceful internal rotation of the thigh in the supine position), the Pace test (abduction of the leg against resistance while sitting) and the Beatty maneuver (active abduction of the thigh on the affected side in the lateral decubitus position) are maneuvers that help in diagnosis. It is known that there is a delay in proximal nerve conduction (H-reflex) on the pathological side compared to the healthy side in the FAIR maneuver on EMG in PS, and it is not a sufficient test for diagnosis alone. Some studies have reported increased piriformis thickness on the pathological side in MRI. None of these clinical and imaging methods are sufficient for diagnosis alone, and today ultrasonography (US) has become one of the most important imaging methods for musculoskeletal clinicians in the diagnosis of PS. Imaging with US and the diagnostic injection test applied to the piriformis muscle with US guidance are quite important for diagnosis. There are a number of studies in the literature evaluating PM with US. These studies have shown that the piriformis muscle thickness and echogenicity increase on the pathological side. However, there is a lack of studies in the literature focusing on the evaluation of the sciatic nerve with US in patients with PS. Our aim in this study is to compare the thickness of the PM and the sciatic nerve by measuring US on both the pathological and painless sides in patients with unilateral hip pain who were diagnosed with PS clinically, to record the variations present in the sciatic nerve, and to determine whether the myofascial pain or the neuropathic component is dominant in the disease.

DETAILED DESCRIPTION:
The sciatic nerve is the largest nerve in the body and is formed by the ventral roots of the lumbosacral plexus (L4-S3), passes through the foramen ischiadicum majus under the piriformis muscle (PM) and enters the gluteal region. It is controversial whether anatomical variations in the sciatic nerve and PM predispose to the development of Piriformis syndrome (PS). The sciatic nerve passes under the PM as a single branch in almost 90% of cases. However, there are some variations where it passes above and through the muscle or divides into tibial and peroneal branches, with one branch passing under the piriformis. There are a number of studies in the literature evaluating the PM with US. These studies have shown that the PM thickness and echogenicity increase on the pathological side. In addition, it has been mentioned that the sciatic nerve has a coarse and blurry image in patients complaining of sciatic pain. In one study, cross-sectional area measurement was performed instead of PM thickness measurement. However, this was criticized in later studies, and it was stated that it was difficult to calculate muscle volume exactly with two-dimensional US due to the irregular shape of the PM, which is anatomically pear-shaped, and that thickness measurement would provide more accurate results instead of cross-sectional area. In the first study in the literature focusing on the sciatic nerve in PS and the neuropathic pain it causes, it was found that the sciatic nerve was significantly enlarged (75%) on the symptomatic side and had decreased echogenicity in some patients when compared to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 70 years with unilateral hip and/or leg pain
* Positive FAIR (flexion, adduction, internal rotation) test
* Tenderness to palpation in the Piriformis muscle

Exclusion Criteria:

* Patients with a history of previous surgery involving the lumbar and/or hip region
* A history of malignancy or infection in the pelvic region
* Body mass index (BMI) Greater than 30 kg/m2
* Psychiatric diseases
* Vascular disease
* Uncontrolled diabetes, hypertension or heart failure,
* Disc pathologies that may cause radiculopathy
* History of rheumatic disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged between 18 and 70 years with unilateral hip and/or leg pain, positive FAIR (flexion, adduction, internal rotation) test, and tenderness to palpation in the PM will be included in our study.
Sampling Method: Probability Sample
Enrollment: 19 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
numeric scale | five months
  Tenderness in the piriformis muscle will be assessed by palpation using the numerical scale (NRS). The numerical scale is a pain score and is evaluated between 0 and 10.
Sciatic nerve thickness (measurement with US) | five months
  Sciatic nerve thickness will be measured with ultrasound on the symptomatic and asymptomatic sides in the same patient.
Piriformis muscle thickness (measurement with US) | five months
  Piriformis muscle thickness will be measured with ultrasound on the symptomatic and asymptomatic sides in the same patient.

CONTACTS AND LOCATIONS:
Overall Officials: Selim Sezikli, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- İstanbul Üniversitesi - Cerrahpasa (IUC), Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No